CLINICAL TRIAL: NCT00005938
Title: A Phase II Study of Intravenous DX-8951f Administered Daily for Five Days Every Three Weeks to Patients With Biliary Tree Cancer (Cholangiocarcinoma and Gallbladder Cancer)
Brief Title: DX-8951f in Treating Patients With Biliary Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067736; DAIICHI-8951A-PRT020; MDA-ID-99379; MSKCC-99110; SACI-IDD-99-31; UCHSC-00892; UTHSC-9905011256
Record Dates: First submitted 2000-07-05; First posted 2004-04-20 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer
Keywords: localized gallbladder cancer; unresectable gallbladder cancer; recurrent gallbladder cancer; localized extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; liver and intrahepatic biliary tract cancer; cholangiocarcinoma of the gallbladder; cholangiocarcinoma of the extrahepatic bile duct; adult primary cholangiocellular carcinoma
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of DX-8951f in treating patients who have biliary cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor activity of DX-8951f in terms of antitumor response, response duration, and survival in patients with biliary tree cancer. II. Evaluate the quantitative and qualitative toxicities of this treatment regimen in this patient population. III. Evaluate the pharmacokinetics of DX-8951 in plasma.

OUTLINE: Patients receive DX-8951f IV over 30 minutes daily for 5 days. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for survival.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed cholangiocarcinoma, bile duct cancer, or gallbladder cancer with or without evidence of unresectable extrahepatic metastasis Previously untreated disease OR Progressive disease after first line chemotherapy Bidimensionally measurable disease by CT scan, chest x-ray, or MRI of the abdomen No known brain metastases

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 2.0 mg/dL Albumin at least 2.8 g/dL SGOT or SGPT no greater than 5 times upper limit of normal (ULN) PT or INR no greater than 1.5 times ULN (if not on Coumadin therapy) Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No active congestive heart failure No uncontrolled angina No myocardial infarction within the past 6 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception before and during study No concurrent serious infection No other life threatening illness No overt psychosis or mental disability that would preclude informed consent No other malignancy within the past 5 years, except: Curatively treated nonmelanomatous skin cancer Carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy and recovered No prior camptothecin analogues No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: At least 4 weeks since prior major surgery and recovered No concurrent surgery Other: No other concurrent anticancer therapy At least 4 weeks since prior investigational drugs No other investigational drugs during or within 4 weeks after final dose of study drug No concurrent drugs that induce or inhibit CYP3A enzyme

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-03; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (5):
- United States (5):
  - University of Colorado Cancer Center, Denver, Colorado
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy & Research Center, San Antonio, Texas